CLINICAL TRIAL: NCT02628483
Title: A Randomized, Double-blind, Parallel Clinical Trial to Compare the Relative Efficacy of Two Triglyceride Forms of Fish Oil, Ultimate Omega®, and a Comparator Product, in Improving Red Blood Cell Fatty Acid Profiles in Healthy Adults (FORCE Study)
Brief Title: A Comparator Trial on the Relative Efficacy of Two Triglyceride Forms of Fish Oil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Pharma, USA (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 1007-008-PRO-040414
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultimate Omega (Experimental): 5 capsules of Ultimate Omega fish oil daily in the morning with food
  Interventions: Dietary Supplement: Fish Oil
- Meg-3 (Active Comparator): 5 capsules of Meg-3 fish oil daily in the morning with food
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Fish Oil — 1000mg fish oil per capsule (325mg EPA + 225mg DHA)
  Other Names: Ultimate Omega
  Arms: Ultimate Omega
Dietary Supplement: Fish Oil — 1000mg fish oil per capsule (300mg EPA + 200mg DHA)
  Other Names: Meg-3
  Arms: Meg-3

SUMMARY:
The health benefits of omega-3 fatty acids have been extensively examined in many published studies, and these benefits have been observed in patients with a diversity of conditions and diseases, including cardiovascular disease (e.g. atrial fibrillation, atherosclerosis, thrombosis, inflammation, sudden cardiac death, etc.), age-related cognitive decline, periodontal disease, rheumatoid arthritis, etc. These fatty acids may also be beneficial to healthy individuals, in terms of preventative health benefits. The balance between omega-6 long chain fatty acids and their omega-3 counterparts is important in health maintenance. An omega-6:omega-3 ratio of 1:1 or 2:1 is recommended for optimal health, yet the average ratio in the North American population is estimated to be as much as 10:1 or even 20:1. A 2014 study of the dietary habits of U.S. adults revealed that, in general, North Americans do not meet the recommended omega-3 fatty acid intake from foods alone. Supplementation may need to be considered, in order to help this population meet their daily needs. Both the Academy of Nutrition and Dietetics and the American Heart Association suggest a prudent approach in recommending an increased intake of omega-3 fatty acids. Although both organisations recommend a preference for obtaining omega-3 fatty acids through fish consumption, both also recognise that supplementation may also be required in order to meet target values, particularly in at-risk populations.

Several omega-3 fish oil supplements exist on the market each with their own ratios of EPA and DHA and are available in varying forms including ethyl ester and high triglyceride forms. Differences in product formulation have been shown to have varying health effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 18 - 35 (inclusive)
* Healthy as determined from medical history
* Non-smoker, or ex-smoker ≥6 months
* Body mass index 18.5 - 24.9 kg/m2
* Female participants of childbearing potential (i.e. not surgically sterilized or post-menopausal greater than one year) must have negative urine pregnancy test and must be using an effective birth control method
* Willing to avoid alcohol consumption for 24 h prior to every clinic visit
* Willing to maintain a stable body weight, activity level and dietary pattern except for use of the study products, as directed
* Willing and able to provide informed written consent

Exclusion Criteria:

* Individuals taking prescription or non-prescription health products that may affect the study endpoint (e.g. corticosteroids, prescription anti-inflammatory drugs, blood lipid-lowering drugs (e.g. statins, fibrates, bile acid exchanger resin, phytosterols, niacin or its analogues, carnitine, etc.) in the previous 6 months
* Individuals taking any supplements with omega-3 fatty acids, phytosterols, polyglucosamines (Chitosan) or other lipid-binding ingredients in the previous 6 months
* Individuals who consume omega-3 fatty acid rich fish (salmon, mackerel, herring) more than twice per month
* Unstable use (initiation or change in dose) of antihypertensive medications or thyroid hormone replacement medications within 3 months prior to visit 1
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 6 months prior to visit 1 and throughout the study
* Pregnancy or lactation, or participant unwilling to take appropriate contraceptives for the duration of the study
* History of blood clotting disorders or use of coagulation-inhibiting drugs (e.g. warfarin)
* Presence of major diseases such as diabetes, gastrointestinal, endocrine, cardiovascular, renal, or liver disease
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.)
* History of cancer (excluding non-melanoma skin cancer and basal cell carcinoma) in past 5 years
* Uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* Abnormal laboratory test results of clinical significance, including, but not limited to, ALT or AST ≥1.5X the upper limit of normal at screening (visit 1)
* Triglycerides ≥400 mg/dL (≥4.52mmol/L) at screening (visit 1)
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Participant has a known allergy or intolerance to fish/fish oil or any of the ingredients in the test products
* Participant is vegan
* Participant is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study, or put the participant at risk
* Participant has taken an investigational medicine or has participated in a research study within 30 days prior to the first study visit

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Red blood cell EPA and DHA | 24 weeks
Phospholipid EPA and DHA | 4 weeks

SECONDARY OUTCOMES:
Red blood cell EPA and DHA | 12 and 16 weeks
Lipid profile | 24 weeks
  Total cholesterol, LDL-C, HDL-C and triglycerides

OTHER OUTCOMES:
Safety Anthropometric Measurements | 4, 12, 16 and 24 weeks
  Blood pressure, Heart rate, Weight and BMI
Safety blood parameters | 24 weeks
  Complete blood count, electrolytes, markers of kidney and liver function
Adverse Events | 24 weeks
  Adverse events over the supplementation period

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No